CLINICAL TRIAL: NCT07058389
Title: Synergy Between Physical Activity and Outdoor Green Environments to Reduce the Intensity of Negative Symptoms in Schizophrenia: a Pilot Study.
Brief Title: Synergy Between Physical Activity and Outdoor Green Environments to Reduce the Intensity of Negative Symptoms in Schizophrenia.
Acronym: SAPIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Jean Monnet University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25CH062; 2025-A00700-49 (Other: ANSM)
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Schizoaffective Disorder
Keywords: Schizophrenia disorders; Mental health; Quality of life; Physical fitness
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INT group (Experimental): 8-week indoor physical activity program (in a gymnasium)
  Interventions: Other: 8-week indoor physical activity program
- EXT group (Experimental): 8-week outdoor physical activity program
  Interventions: Other: 8-week outdoor physical activity program
- TEM group (No Intervention): Without physical activiy program (no change in routine)

INTERVENTIONS:
Other: 8-week outdoor physical activity program — EXT group will perform aerobic and resistance exercises with a coach in adapted physical activities on a green environment in a parc.
  Sessions will be typically composed as follows:
  * Warm-up (20 min)
  * Aerobic exercise (30 min) at RPE 4 to 7 on the Borg scale
  * Muscular strengthening (25 min) at RPE 4 to 7 on the Borg scale
  * Cool-down, stretching and balance (15 min) EXR group will train for 8 weeks, twice a week for 1h30, following WHO recommendation.
  Arms: EXT group
Other: 8-week indoor physical activity program — INT group will perform aerobic and resistance exercises with a coach in adapted physical activities, inside a conventional gym.
  Sessions will be typically composed as follows:
  * Warm-up (20 min)
  * Aerobic exercise (30 min) at RPE 4 to 7 on the Borg scale
  * Muscular strengthening (25 min) at RPE 4 to 7 on the Borg scale
  * Cool-down, stretching and balance (15 min) INT group will train for 8 weeks, twice a week for 1h30, following WHO recommendation.
  Arms: INT group

SUMMARY:
Physical activity appears to be a novel and original adjunctive therapeutic approach in the management of patients with schizophrenia. It may help reduce schizophrenic symptoms, act as a pro-cognitive therapy, improve quality of life, and reduce cardiovascular comorbidities. Moreover, some evidence suggests that physical activity practiced in a natural environment has even more positive effects on mental health compared to physical activity carried out indoors or in urban settings. Indeed, greater exposure to greenery is associated with a better perception of general health and with reduced levels of cortisol, anxiety, and depression. No study has yet attempted to examine the impact of physical activity in green (outdoor) spaces compared to indoor physical activity on the negative symptoms of patients suffering from schizophrenia. The aim of this study is therefore to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia, aged 18 to 55 years
* Having persistent negative symptoms (SNS), negative symptoms self-assessment scale > 7
* Regularly monitored in the psychiatry department.
* Have no medical contraindications to physical activity
* Subject affiliated with or entitled to a social security system.
* Subject having received informed information about the study and having co-signed, with the investigator, consent to participate in the study.
* Male or female.

Exclusion Criteria:

* Patient unsuitable for study in the opinion of the investigator
* Any subject with chronic joint pathologies (example: repeated sprains, patellar or ligament problems) or cardiac pathologies.
* Any subject presenting chronic or central neurological pathologies.
* Any subject deprived of liberty or subject to legal protection
* Excessive consumption of alcohol (> 14 glasses per week) or caffeinated drinks (> 400 mg of coffee per day).
* Pregnant women.
* Subject unable to understand the purpose and conditions of the study, unable to give consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Self-evaluation of negative symptoms (SNS) questionnaire | Weeks 2, 10 and 22
  The primary outcome will be the evolution of negative symtoms, assessed using the Self-evaluation of negative symptoms (SNS) questionnaire. The total SNS score ranges from 0 to 40, where higher scores indicate greater severity of negative symptoms.

SECONDARY OUTCOMES:
Clinical global Impression (CGI) scale | Weeks 2, 10 and 22
  The patient's overall symptomatology and functioning will be assessed by the Clinical global Impression (CGI) scale. The CGI scale is assessed on a 7-point scale, with the severity of illness rated from 1 (normal) to 7 (very seriously ill). CGI scores range from 1 (much improved) to 7 (much worse).
Personal and social performance (PSP) scale | Weeks 2, 10 and 22
  The patient's overall symptomatology and functioning will be assessed by the Personal and social performance (PSP) scale. Higher scores indicate higher levels of perceived stress.
Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS) | Weeks 2, 10 and 22.
  Cognitive disorders reported will be assessed using the French version of the Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS). The total score (range 0-84) is calculated as the sum of all items, with higher scores reflecting a greater Self-Appraisals of Cognitive Deficits.
VO2 max | Weeks 2, 10 and 22.
  VO2 max will be estimated on the basis of heart rate measured during a submaximal test on an ergonomic bicycle.
Maximum force | Weeks 2, 10 and 22.
  The maximum force produced by the knee extensors will be measured on a dynamometer.
Flexibility | Weeks 2, 10 and 22.
  Flexibility of the posterior chain will be measured with the sit and reach test.
Spatio-temporal coordination | Weeks 2, 10 and 22.
  Spatio-temporal coordination will be assessed by measuring individual reaction times.
Balance | Weeks 2, 10 and 22.
  Balance will be tested by stabilometry on a Winposturo force platform.
IPAQ questionnaire | Weeks 2, 10 and 22.
  The level of sedentariness will be measured by the IPAQ questionnaire. This questionnaire classifies the subject according to 3 levels of activity: inactive, moderate, high.

CONTACTS AND LOCATIONS:
Overall Officials: Medhi HOUSNI, Md, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France, France

IPD SHARING:
Plan to Share IPD: No